CLINICAL TRIAL: NCT00900523
Title: Urine Prostaglandin-M(PGE-M) in Ovarian Cancer
Brief Title: Prostaglandin Metabolite in Urine Samples From Patients With Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Marta Crispens, MD, Associate Professor; Gynecological Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC GYN 0648; VU-VICC-GYN-0648; VU-VICC-IRB-060680
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Ovarian Cancer
Keywords: recurrent ovarian epithelial cancer; stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — 7-hydroxy-5,11-dioxotetranorprostane-1,16-dioic acid; Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Known or suspected ovarian cancer: Women who have a diagnosis of ovarian cancer or who are suspected of having ovarian cancer
  Interventions: Genetic: protein expression analysis; Other: immunohistochemistry

INTERVENTIONS:
Genetic: protein expression analysis — protein expression analysis
  Other Names: protein expression analysis for PGE-M
Other: immunohistochemistry — immunohistochemical staining of tumor tissue to measure COX-1 and COX-2 levels
  Other Names: immunohistochemistry staining methods

SUMMARY:
RATIONALE: Measuring the amount of prostaglandin metabolite in urine samples and studying tissue samples in the laboratory from patients with ovarian cancer may help doctors identify and learn more about biomarkers related to ovarian cancer and may help the study of cancer in the future.

PURPOSE: This laboratory study is measuring the amount of prostaglandin metabolite in urine samples from patients with ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the level of prostaglandin E_2 metabolite (PGE-M) in 24-hour urine samples collected prior to surgery or chemotherapy from patients with ovarian cancer.
* Determine cyclooxygenase-1 (COX-1) and cyclooxygenase-2 (COX-2) expression by western blot and immunohistochemistry (IHC) in ovarian tumor tissue samples and matched normal ovarian tissue samples, if available, from these patients.
* Correlate urine PGE-M levels with corresponding tissue COX-1 and COX-2 levels in urine and tissue samples from these patients.

OUTLINE: This is a pilot study.

Patients submit 24-hour urine specimens prior to surgery for evaluation of urinary levels of prostaglandin E_2 metabolite (PGE-M).

Patients also undergo assessment of tissue obtained at the time of surgery, including ovarian tumor tissue, normal surface ovarian epithelium tissue (if available), and fixed tissue embedded in a paraffin block. Tissue samples are analyzed by western blot and IHC for cyclooxygenase-1 and cyclooxygenase-2 expression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of known or suspected ovarian cancer
* Age greater than 17 years

Exclusion Criteria:

* Pregnant or nursing
* Taking steroids or non-steroidal anti-inflammatory drugs (NSAIDs) on a regular basis.

PRIOR CONCURRENT THERAPY:

* No concurrent chronic use of steroids or NSAIDs

Min Age: 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with known or suspected ovarian cancer who are greater than 17 years in age.
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2006-11; Primary Completion 2007-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Prostaglandin E2 metabolite (PGE-M) levels in 24-hour urine samples | Pre-surgical or chemotherapeutic treatment, over a 24-hour duration
  Patients will be collect their urine for 24 hours before they undergo any surgery or chemotherapy. Researchers will measure the amount of PGE-M in the urine.

SECONDARY OUTCOMES:
COX-1 and COX-2 expression in ovarian tumor tissue and non-malignant tissue | Day of surgery
  COX-1 and COX-2 expression will be measured in samples of patients' malignant ovarian samples and matched non-malignant samples (the latter if available).
Correlation of urine PGE-M levels with tissue COX-1 and COX-2 levels | After patients' surgery
  Patients' levels of urine PGE-M will be compared and contrasted with their levels of COX-1 and COX-2 in ovarian tumor tissue

CONTACTS AND LOCATIONS:
Overall Officials: Marta Crispens, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center